CLINICAL TRIAL: NCT05896423
Title: Increasing PrEP Awareness and Demand Among Black Cisgender Women
Acronym: IPAD-BCW
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Howard Brown Health Center (Other); Planned Parenthood of Illinois (Unknown); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Maria Pyra, Assistant Professor, Northwestern University
Other Study IDs: STU00218358; P30AI117943 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: HIV; PrEP
Keywords: cis women; Black women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBH cohort: Rates of PrEP initiation among Black cis women at an FQHC, before and after the PrEP materials are used
  Interventions: Behavioral: PrEP awareness materials
- PPIL cohort: Rates of PrEP initiation among Black cis woman at a family planning clinic, before and after the PrEP materials are used

INTERVENTIONS:
Behavioral: PrEP awareness materials — Community-designed PrEP awareness materials - developed in the formative portion of this study
  Groups: HBH cohort

SUMMARY:
This study will develop HIV pre-exposure prophylaxis (PrEP) awareness materials for and with Black cis women and gather feedback on the usefulness of these materials at health care sites. The investigators will also use electronic medical records (EMR) to compare the number of Black cis women who initiate PrEP before and after the awareness materials are piloted, at the two partner research sites, Howard Brown Health and Planned Parenthood of IL. Additional federally qualified health centers and family planning clinics will review the materials and complete a survey on acceptability.

DETAILED DESCRIPTION:
Aim 1. Develop digital PrEP awareness materials to engage Black cis women. Using Human Centered Design and guided by (capability, opportunity, motivation, behavior; Theoretical Domains Framework)COM-B+TDF as a behavior change theory, the investigators will conduct 5 focus groups across two clinical sites with Black cis women ages 16 to 40 from high HIV-prevalence areas of Chicago (n=120 participants). This iterative process, in collaboration with the HBH communications team and led by an experienced human centered design (HCD) researcher, will lead to the development of digital PrEP awareness materials that will be piloted online. Through qualitative analysis of the focus groups, the investigators will generate knowledge regarding how TDF can be used to understand HIV prevention in this population.

Aim 2. Assess acceptability and feasibility of the PrEP awareness materials in new FQHC & family planning clinics in Ending the HIV Epidemic (EHE) jurisdictions. Guided by implementation science frameworks and tools, the investigators will develop a toolkit and survey to accompany pilot distribution. The toolkit will provide guidance on using and adapting the awareness materials, based in the behavior change knowledge developed in aim 1. The survey will assess the acceptability, appropriateness, and feasibility of using the awareness materials, to prepare for further assessment and dissemination. The awareness materials, toolkit, and survey will be distributed locally and outside of Illinois, through Federally Qualified Health Centers and Planned Parenthood networks, as well as the Third Coast Center for AIDS Research (CFAR) and Getting to Zero networks, with a target of 20 online surveys collected.

ELIGIBILITY:
Inclusion Criteria:

* identify as cis women
* identify as Black or African-American
* self-report not living with HIV
* reside in a high HIV incidence neighborhood in Chicago
* aged 16 to 40, inclusive
* able to speak English.

Exclusion Criteria:

* Unable to provide consent

Ages: 16 Months to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender women
Study Population: Black cis women living in high HIV incidence areas of Chicago
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Black cis women initiating HIV PrEP | ~June 2023-June 2024
  Number of Black cis women at each clinic with first prescription for any form of HIV PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pyra, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Planned Parenthood of Illinois, Chicago, Illinois
  - Howard Brown Health, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be available